CLINICAL TRIAL: NCT05124743
Title: HLA Typing and Tumor Neoantigen Identification for a Phase I/II Study of Autologous T-Cell Receptor-Engineered T Cells (TCR-T) Reactive Against Cancer-specific Mutations in Subjects With Solid Tumors
Brief Title: HLA Typing & Tumor Neoantigen Identification for Phase I/II Study of Autologous TCR-T Cells in Subjects With Solid Tumors
Status: Terminated | Type: Observational
Why Stopped: TCR001-002 protocol was combined with TCR001-201 protocol, which was terminated due to business decisions.
Sponsor: Alaunos Therapeutics (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: TCR001-002
Record Dates: First submitted 2021-10-18; First posted 2021-11-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Colo-rectal Cancer; Cholangiocarcinoma; Non-small Cell Lung Cancer; Pancreas Cancer
Keywords: TCR, solid tumor, TCR-T, neoantigen, Alaunos
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Colonic Neoplasms; Cholangiocarcinoma; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a data collection study, also referred to as a "screening" study; no investigational or standard therapy will be administered as part of this study. In order to identify subjects for the Phase I/II study, TCR001-201, patients with following histologically confirmed tumor types will be initially screened in this protocol for their somatic mutation and HLA type:

* Gynecologic cancer (ovarian or endometrial)
* Colorectal cancer
* Pancreatic cancer
* Non-small cell lung cancer (NSCLC). NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma or adenocarcinomas
* Cholangiocarcinoma Subjects' somatic mutation(s) and HLA type restriction combination will be examined against Alaunos Therapeutics Inc.'s (Alaunos) TCR library to determine if a TCR match is available for that subject. Subjects without a match will be discontinued from this protocol.

Subjects with a TCR match in the Alaunos TCR library will continue to be followed on this protocol and their clinical status will be monitored on an ongoing basis for eligibility, i.e., for progressive or recurrent disease, to enroll and receive TCR-T cell therapy on the Phase I/II study. Subjects will complete participation on this protocol when the subject enrolls on the Phase I/II study or if the subject dies.

DETAILED DESCRIPTION:
This protocol will be used to perform and/or collect results from genetic mutation testing (e.g., Oncomine™ or similar genomic test performed at a CLIA-certified laboratory) and high resolution, human leukocyte antigen (HLA) class I and II typing from a CLIA-certified laboratory. This protocol will also collect subject clinical baseline characteristics, demographics, and cancer history. This protocol will be used to monitor subject disease status to identify candidates for enrollment onto the Phase I/II study as patients must have progressive or recurrent disease to be enrolled onto that protocol.

The subject's somatic mutation(s) and HLA type restriction combination will be examined against Alaunos' TCR library to determine if a TCR is available for that subject. Subjects without a TCR match will be discontinued from this protocol. If the subject's somatic mutation and HLA type restriction combination matched TCR is added to the Alaunos TCR library after the subject discontinues, the investigator may contact the subject to be re-screened for the study.

Subjects with a TCR match in the Alaunos TCR library will continue to be followed on this protocol and their clinical status will be monitored on an ongoing basis for eligibility, particularly progressive or recurrent disease, to enroll and receive TCR-T cell therapy on the Phase I/II study. Clinical status will be collected at enrollment and approximately every 3 months in conjunction with subjects' regularly scheduled standard of care visits. Subjects with a TCR match will complete participation on this protocol once they enroll in the Phase I/II study or if the subject dies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have previously received at least one line of standard systemic therapy for their advanced/metastatic cancer, and have either progressed, recurred or were intolerant to the previous treatment for one of the following cancer types:

   1. Gynecologic cancer (ovarian and endometrial)
   2. Colorectal cancer
   3. Pancreatic cancer
   4. Non-small cell lung cancer (NSCLC), NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma or adenocarcinomas
   5. Cholangiocarcinoma
2. Patients with previous tumor genomic testing performed at a CLIA-certified laboratory must be willing to disclose results. Patients that do not have previous tumor genomic testing must have a planned biopsy or resection as part of their standard of care (or archived tumor tissue available for genomic testing) or must provide a blood sample for circulating tumor DNA (liquid biopsy) testing. If prior genomic testing results or archival biopsy with sufficient tumor tissue are older than 6 months, a new tumor biopsy is required if being performed as standard-of-care. If re-biopsy is not feasible, a liquid biopsy must be performed to confirm previous test results.
3. Patients with previous high resolution, human leukocyte antigen (HLA) class I and II typing from a CLIA certified laboratory must be willing to disclose results. Patients that do not have previous typing results must be willing to provide a blood sample for this testing.
4. Patients must be able to provide written informed consent.
5. Patients must be age greater than or equal to 18 years.
6. Patients must have a clinical performance status of Eastern Cooperative Oncology Group (ECOG) of 0 or 1. Patients with an ECOG of 2 may be acceptable with Medical Monitor approval.

Exclusion Criteria:

1. Any other unstable or clinically significant medical condition that would, in the opinion of the Principal Investigator (PI) in consultation as warranted with medical monitor, result in risks to safety of a subject and/or their compliance with the protocol. Examples include, but are not limited to, a history of myocarditis or congestive heart failure (New York Heart Association functional Class III or IV), unstable angina, serious uncontrolled cardiac arrythmia, myocardial infarction within 6 months of screening, active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring chronic treatment with systemic steroids, uncontrolled asthma, or colitis.
2. Any form of primary immunodeficiency (such as severe combined immunodeficiency disease).
3. Has another concurrent clinically active hematologic malignancy or solid tumor malignancy requiring treatment, except for non-melanoma cancers of the skin, carcinoma in situ of the cervix, or non-metastatic prostate cancer.
4. Has a history of a bleeding disorder or unexplained major bleeding diathesis or is currently receiving chronic anticoagulation therapy.
5. Has received any type of organ transplant in the past 12 months.
6. Has undergone xenotransplantation at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously received at least one line of standard systemic therapy for their advanced/metastatic cancer, and have either progressed, recurred or were intolerant to the previous treatment for one of the following cancer types:
  1. Gynecologic cancer (ovarian or endometrial)
  2. Colorectal cancer
  3. Pancreatic cancer
  4. Non-small cell lung cancer (NSCLC); NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma or adenocarcinomas
  5. Cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Positive for Human Leukocyte Antigen (HLA)-A*02 | Screening Visit
  A blood sample was collected from each consented participant to determine their human leukocyte antigen (HLA) haplotype. This measure reports the number of subjects identified as positive for the HLA-A*02 allele, which was a key eligibility criterion for potential enrollment into the subsequent treatment protocol (TCR001-201)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No